CLINICAL TRIAL: NCT01617798
Title: Stop Hypernatremia, Use Metolazone for Aggressive, Controlled, Effective Diuresis
Brief Title: Stop Hypernatremia, Use Metolazone, for Aggressive, Controlled, Effective Diuresis
Acronym: SHUM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator departed organization
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Gold, Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007857
Record Dates: First submitted 2012-06-01; First posted 2012-06-12 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Failure; Volume Overload; Hypernatremia
MeSH Terms: conditions — Respiratory Insufficiency; Edema; Hypernatremia | interventions — Furosemide; Single Person; Metolazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control-- furosemide (lasix) only (Placebo Comparator): Control arm receives standard of care diuresis with furosemide(lasix)only. The treatment team will decide the dosing of furosemide (lasix).
  No actual placebo is administered.
  Interventions: Drug: Placebo Comparator: Control-- furosemide (lasix) only
- Study Arm (Active Comparator): Study arm receives evolving standard of care diuresis with furosemide and metolazone.
  Interventions: Drug: Supplemental metolazone diuresis

INTERVENTIONS:
Drug: Supplemental metolazone diuresis — Patients in the Study Arm will receive supplemental diuresis with metolazone 2.5 mg per dobhoff tube twice daily, in addition to furosemide as the primary team sees fit.
  Other Names: furosemide, lasix
  Arms: Study Arm
Drug: Placebo Comparator: Control-- furosemide (lasix) only — Control arm will receive furosemide as monotherapy for diuresis
  Other Names: furosemide, lasix, metolazone
  Arms: Control-- furosemide (lasix) only

SUMMARY:
Patients who are on mechanical ventilation in an intensive care unit often require diursis as part of their pre-extubation regimen. The drug of choice for diuresis has traditionally been furosemide. However, this drug cause hypernatremia (a rise in serum sodium) in a significant proportion of patients. Hypernatremia is traditionally treated by providing free water supplementation to the patient. This strategy creates a vicious and unproductive cycle of giving free water, and then diuresing it off. We propose a strategy for breaking this cycle by using a second diuretic-- metolazone-- which has a tendency to rid the body of more sodium, thereby minimizing hypernatremia.

DETAILED DESCRIPTION:
Mechanical ventilation is a mainstay of Intensive Care. Weaning from mechanical ventilation remains a significant issue in Intensive Care Unit (ICU) care worldwide. It is well established that a strategy of diuresis with negative fluid balance shortens the duration of mechanical ventilation in both acute lung injury and cardiogenic pulmonary edema patients. Despite publication of at least one formalized but complex evidence-based conservative fluid strategy, there is no practical, uniformly implemented protocol for setting or achieving volume status targets. The default approach at many hospitals involves using ad hoc doses (either intermittent or continuous) of a loop diuretic (usually furosemide) with instructions to monitor fluid balance and follow electrolytes in an attempt to reach arbitrary target volume diuresis. Moreover, there are barriers to achieving any particular target, including pre-existing renal failure/diuretic resistance, diuretic-induced creatinine elevation, acquired diuretic resistance, hypotension from volume loss, and electrolyte derangements including hypokalemia and hypernatremia. Strategies exist for preventing or treating the above complications but there is presently no accepted standard for preventing or treating diuretic-induced hypernatremia. In fact, the standard current intervention is to replace the free water deficit that may be induced by the loop diuretic, while simultaneously perpetuating the free water deficit by continuing to administer the causative loop diuretic. This approach is circular and does not effectuate the desired negative fluid balance. We will address the lack of an accepted prevention strategy using a randomized controlled clinical trial in ICU patients with the following specific aims:

1. Conduct a randomized, pilot trial of standard versus metolazone supplemented diuresis in ICU patients with the primary outcome of improved negative fluid balance.
2. Assess secondary outcomes including time to extubation, exacerbation of renal failure, and incidence of electrolyte derrangements in the treatment and control arms.
3. Track whether initial hypernatremia within the control group is a risk factor for poor diuresis with furosemide, and whether it delays extubation.

The anticipated benefits of our proposed intervention involve fundamental ICU and patient care quality measures: avoiding the pitfalls of hypernatremia and diuretic resistance should lead to more effective diuresis, which should in turn lead to a more negative fluid balance, earlier liberation from the ventilator, and a shorter length of stay in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who are intubated and slated for diuresis in anticipation of extubation.
* Patients must be hypernatremic (Na > 140 mEq/L) at the time diuresis is initiated or become hypernatremic over the course of receiving loop diuretics in anticipation of extubation.
* GFR > 30 ml/min [as calculated by the MedCalc MDRD formula {GFR = 170 x PCr - 0.999 x Age - 0.176 x BUN - 0.170 x Albumin0.318 x 0.762 (for women) x 1.180 (for blacks)} ]

Exclusion Criteria:

* History of allergy to furosemide or any thiazide diuretic
* Inability to place enteral access
* Moribund status

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Fluid balance | 24, 36, 48, and 72 hours after either protocol is initiated
  Differences in fluid balance (total net liters negative from the time diuresis is initiated) between the study group and control group at the following intervals: 24, 36, 48, and 72 hours after either protocol is initiated.

SECONDARY OUTCOMES:
Serum sodium | Continuous for 72 hours
  Number patients whose Na remains below 145 (meq/L) during the period of diuresis; versus the number of patients whose sodium exceeds 145 (meq/L) and require free water replacement.
Hyponatremia | Continuous for up to 72 hours
  Number of patients who develop hyponatremia (Na < 136 meq/L)
Time to extubation | Unitl the patient is actually extubated, undergoes tracheostomy, or expires.
  Time in hours from initiation of protocol to extubation (difference between study group and control group
Acute Kidney Injury | Continuous for the first 72 hours
  Number of patients who develop acute kidney injury (increase in creatinine by more than 25%)

CONTACTS AND LOCATIONS:
Overall Officials: David Steiger, JD MD, Principal Investigator — Oregon Health and Science University; Dan Hagg, MS MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States